CLINICAL TRIAL: NCT05599269
Title: Retrospective Clinical Evaluation of Nano-hybrid-composite Denture Teeth SR Phonares II
Brief Title: Retrospective Clinical Evaluation of Nano-hybrid-composite Denture Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ivoclar Vivadent AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LL5267725
Record Dates: First submitted 2022-10-20; First posted 2022-10-31 (Actual); Results first posted 2025-03-28 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Edentulous Mouth; Dental Prosthesis Failure
MeSH Terms: conditions — Mouth, Edentulous

STUDY DESIGN:
Intervention Model Description: retrospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Examination of dentures with SR Phonares II teeth (Other)
  Interventions: Device: Examination of dentures with SR Phonares II teeth

INTERVENTIONS:
Device: Examination of dentures with SR Phonares II teeth — The intraoral situation will be examined similar to a standard dental examination. The dentures are then removed, cleaned and examined extraoral. Pictures and an impression of the dentures are taken.

SUMMARY:
This retrospective study investigates the longevity of dentures with SR Phonares II teeth after a wearing period of more than 10 years.

The primary objective is to assess the survival rate of dentures with SR Phonares II teeth after more than 10 years. The secondary objectives asses the quality of the dentures concerning aesthetic, functional and biological properties.

ELIGIBILITY:
Inclusion Criteria:

* informed consent signed and understood by the subject
* partial or full denture with SR Phonares II teeth
* dentures delivered in the internal clinic between August 2010 and August 2012
* to be able to visit the internal clinic (Exception: Patients with limited mobility are also included if another person can carry the dentures to the internal clinic of Ivoclar Vivadent AG for the examination.)

Exclusion Criteria:

* patient does not wear the dentures regularly
* health status (physical and mental) does not allow participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-11-18 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2023-04-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ivoclar Vivadent AG, Schaan, Liechtenstein

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Examination of dentures with SR Phonares II teeth
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Examination of dentures with SR Phonares II teeth
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 16
Age, Continuous [Mean (Full Range); unit: years] | 77 [61 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 17
Region of Enrollment [Number; unit: participants]
  Liechtenstein | 17

OUTCOME MEASURES:

1. Primary Outcome: Survival Rate of Dentures With SR Phonares II Teeth
Description: After a wearing time of 10 years dentures with SR Phonares II teeth were examined by a dentist
Time Frame: 10 years
Measure: Count of Participants; unit: Participants
Arm/Group | Examination of dentures with SR Phonares II teeth
Number analyzed (Participants) | 17
Participants | 17

2. Secondary Outcome: Quality of the Dentures Concerning Aesthetic, Functional and Biological Properties
Description: After a wearing time of 10 years dentures with SR Phonares II teeth were evaluated by a dentist according to adopted FDI criteria.
  Aesthetic properties (surface luster, surface staining, plaque accumulation, color match (to a reference), functional properties (fracture of material, marginal adaption, occlusal contour and wear, patient's view (evaluated during discussion) and biological properties (adjacent mucosa, oral health) were eveluated according the following FDI grades:
  * FDI grade 1: clinically excellent
  * FDI grade 2: clinically good
  * FDI grade 3: clinically satisfactory
  * FDI grade 4: clinically unsatisfactory
Time Frame: 10 years
Population: As only the denture was made available for some examinations in the clinical investigation, it was not possible to examine the oral health of these patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Examination of dentures with SR Phonares II teeth
Number analyzed (Participants) | 17
Participants
  surface lustre teeth: Grade 1 | 2
  surface lustre teeth: Grade 3 | 0
  surface lustre teeth: Grade 2 | 15
  surface lustre teeth: Grade 4 | 0
  staining teeth: Grade 1 | 17
  staining teeth: Grade 4 | 0
  staining teeth: Grade 3 | 0
  staining teeth: Grade 2 | 0
  plaque accumulation: Grade 2 | 16
  plaque accumulation: Grade 4 | 0
  plaque accumulation: Grade 1 | 1
  plaque accumulation: Grade 3 | 0
  color match: Grade 1 | 17
  color match: Grade 2 | 0
  color match: Grade 3 | 0
  color match: Grade 4 | 0
  fracture: Grade 4 | 0
  fracture: Grade 2 | 2
  fracture: Grade 1 | 10
  fracture: Grade 3 | 5
  marginal adaptation: Grade 2 | 4
  marginal adaptation: Grade 1 | 12
  marginal adaptation: Grade 4 | 0
  marginal adaptation: Grade 3 | 1
  occlusal contour/wear: Grade 3 | 13
  occlusal contour/wear: Grade 1 | 1
  occlusal contour/wear: Grade 2 | 3
  occlusal contour/wear: Grade 4 | 0
  patients view: number analyzed (Participants) | 16
  patients view: Grade 2 | 0
  patients view: Grade 1 | 16
  patients view: Grade 3 | 0
  patients view: Grade 4 | 0
  adjacent mucosa: number analyzed (Participants) | 15
  adjacent mucosa: Grade 4 | 0
  adjacent mucosa: Grade 1 | 15
  adjacent mucosa: Grade 2 | 0
  adjacent mucosa: Grade 3 | 0
  oral health: number analyzed (Participants) | 15
  oral health: Grade 3 | 0
  oral health: Grade 1 | 14
  oral health: Grade 2 | 0
  oral health: Grade 4 | 1

ADVERSE EVENTS:
Time Frame: retrospective study after 10 years of dentures wear, participants assessed for a maximum of 90 minutes
Description: As it's a retrospective study and patients were examined after 10 years in one recall, it's not possible to define a time frame over which adverse event data were collected. Recall takes a maximum of 90 minutes for each patient.
Arm/Group | Examination of dentures with SR Phonares II teeth
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-19): https://cdn.clinicaltrials.gov/large-docs/69/NCT05599269/Prot_SAP_001.pdf